CLINICAL TRIAL: NCT04609306
Title: How Does Hydrogen Peroxide Application to the Wound Following Surgical Incision Affect C. Acnes Cultures in Primary Shoulder Arthroplasty?
Brief Title: Hydrogen Peroxide to the Wound Following Surgical Incision Affecting Cultures in Primary Shoulder Arthroplast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202002655; OCR39759 (Other: UF OnCore)
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Primary Anatomic or Reverse Total Shoulder Arthroplasty

STUDY DESIGN:
Intervention Model Description: Two group parallel study
Who Masked: Participant
Masking Description: Subjects will then be randomized 1:1 into Experimental or Control cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subjects getting 3% H2O2 applied to the incision (Experimental): For the experimental cohort, a lap sponge soaked in 3% H2O2 will be applied to the incision and allowed to sit for 3 minutes. Following the 3 minutes, the sponge will be removed, the wound will be flushed with 100 mL of normal saline, and the exposed dermis will be swabbed and sent for culture.
  Interventions: Other: H2O2 application to incision
- Subjects not getting 3% H2O2 applied to the incision (No Intervention): In the control cohort, the dermis will be swabbed and sent for culture immediately after the skin incision is made and the knife is removed from the field.

INTERVENTIONS:
Other: H2O2 application to incision — A lap sponge soaked in 3% H2O2 will be applied to the incision and allowed to sit for 3 minutes.
  Arms: Subjects getting 3% H2O2 applied to the incision

SUMMARY:
Cutibacterium acnes has been the focus of much recent shoulder literature, as it has been found to be both a common cause of periprosthetic joint infection as well as a common contaminant in shoulder surgery. Standard skin preparations have been found to be ineffective at eradicating C. acnes colonization on the skin and deep dermis of patients undergoing surgery. Recent literature has shown that skin preparation with 3% hydrogen peroxide solution is effective for decreasing the rate of cultures positive for C. acnes in both dermal and deep cultures; however, a positive rate of 10%-17% has still been reported despite this skin preparations. The current theory is that standard skin preparation does not remove C. acnes from the deep dermis which subsequently contaminates the deep tissue. We hypothesize that application of 3% hydrogen peroxide to the deep dermal layer immediately following the skin incision will even further decrease the rate of C. acnes contamination during surgery.

DETAILED DESCRIPTION:
Over 50,000 people in the United States have shoulder replacement surgery each year. Of these, it is reported that 0.4%-2.9% of anatomic total shoulder arthroplasties (aTSA) and 1-10% of reverse shoulder arthroplasties (rTSA) are complicated by periprosthetic joint infection (PJI).

Cutibacterium Acnes (C. acnes), an indolent organism found on the skin and in the sebaceous glands around the shoulder and back, makes the diagnosis of shoulder PJI particularly challenging. Multiple studies have shown that C. acnes can be isolated from deep cultures in up to 40% of patients without prior surgery undergoing primary total shoulder arthroplasty, although whether this indicates actual colonization of the joint or contamination is an area of debate.

A recent development in shoulder surgery is the use of hydrogen peroxide to decrease the C. acnes load in the deep dermis sebaceous glands, with the hope that this will prevent contamination of the joint during shoulder joint replacement surgery. Application of a widely commercially-available 3% topical Hydrogen peroxide in water solution in vitro has been found to completely eradicate C. acnes growth within 5 minutes and has been shown in clinical trials when used as part of the skin preparation to decrease the rate of positive cultures for C. acnes from 35% to 10% for deep cultures and from 34% to 17% for superficial dermal cultures. While these results show marked improvement compared to standard skin preparations, the 17% with positive dermal cultures is still concerning given the significant morbidity associated with a PJI.

Our hypothesis is that an additional application of hydrogen peroxide to the dermis itself, immediately following the skin incision, will be even more effective at eradicating this potential source of contamination deep in the joint.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, age 40-90
* Undergoing primary anatomic or reverse total shoulder arthroplasty for glenohumeral osteoarthritis or rotator cuff arthropathy

Exclusion Criteria:

* Female patients
* Patients under 40 years or over 90 years of age
* Diagnosis other than glenohumeral osteoarthritis or rotator cuff arthropathy
* Prior arthroscopic or open shoulder surgery on the ipsilateral shoulder
* Prior diagnosis of septic shoulder of the ipsilateral shoulder
* Corticosteroid injection within 3 months of the procedure
* Recently on antibiotics (within 2 weeks) prior to surgery

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 36 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wright, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Getting 3% H2O2 Applied to the Incision | Subjects Not Getting 3% H2O2 Applied to the Incision
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Getting 3% H2O2 Applied to the Incision | Subjects Not Getting 3% H2O2 Applied to the Incision | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Full Range); unit: years] | 67.8 [55 to 81] | 71.8 [60 to 90] | 69.8 [55 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 17 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Positive vs Negative Culture's Based on Skin Prep Method
Description: Following our standard protocols for skin preparation (which includes an application of 3% H2O2, alcohol, and then Chloraprep in sequence) and draping (with Ioban applied over the skin), we will start the procedure as normal. The skin incision will be made in standard fashion, and the knife used will be removed from the surgical field. For the experimental cohort, a lap sponge soaked in 3% H2O2 will be applied to the incision and allowed to sit for 3 minutes. Following the 3 minutes, the sponge will be removed, the wound will be flushed with 100 mL of normal saline, and the exposed dermis will be swabbed and sent for culture. In the control cohort, the dermis will be swabbed and sent for culture immediately after the skin incision is made and the knife is removed from the field.
Time Frame: 3 minutes prior to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Getting 3% H2O2 Applied to the Incision | Subjects Not Getting 3% H2O2 Applied to the Incision
Number analyzed (Participants) | 18 | 17
Participants
  Number of positve cultures | 6 | 6
  Number of negative cultures | 12 | 11

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Subjects Getting 3% H2O2 Applied to the Incision | Subjects Not Getting 3% H2O2 Applied to the Incision
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04609306/Prot_SAP_000.pdf